CLINICAL TRIAL: NCT03951610
Title: A Dispensing Clinical Trial of Invigor 1 Daily Disposable Lens Against Clariti 1-day Lens
Brief Title: A Dispensing Comparison of a Test Daily 1 Day Lens Against a Control 1 Day Lens.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-19-01
Record Dates: First submitted 2019-03-11; First posted 2019-05-15 (Actual); Results first posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: This will be a, prospective, double-masked, randomized, bilateral, 1 week cross-over, dispensing study
Who Masked: Participant, Investigator
Masking Description: Double (participant and investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Test lens (Experimental): Subjects wearing the test lens for one week, either randomized as the first or second pair.
  Interventions: Device: Test lens; Device: Control lens
- Control lens (Active Comparator): Subjects wearing the control lens for one week, either randomized as the first or second pair.
  Interventions: Device: Test lens; Device: Control lens

INTERVENTIONS:
Device: Test lens — contact lens
  Other Names: Invigor I DD lens; Somofilcon A 1 day Test
Device: Control lens — contact lens
  Other Names: Clariti 1-day; Somofilcon A 1 day control

SUMMARY:
The purpose of this study is to compare the dispensing performance of somofilcon A test 1 day contact lens against somofilcon A control 1 day contact lens.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the clinical performance of a silicone-hydrogel test contact lens compared to the commercially available silicone-hydrogel (control) contact lens when worn over one week for each lens type in a randomized, bilateral, cross-over, dispensing study on a daily disposable basis.

ELIGIBILITY:
Inclusion Criteria:

* Has had a self-reported oculo-visual examination in the last two years.
* Is at least 18 years of age and has full legal capacity to volunteer.
* Has read and understood the information consent letter.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Is correctable to a visual acuity of 20/40 or better (in each eye) with their habitual vision correction or 20/20 best-corrected.
* Currently wears soft contact lenses (average wearing of 8 hours/day and 5 days/week) without the need of using rewetting drops
* Requires spectacle lens spherical powers between -1.00 to -5.75 diopters sphere (0.25D steps).
* Has no more than 0.75 diopters of refractive astigmatism.
* Has clear corneas and no active ocular disease.
* Has not worn lenses for at least 12 hours before the examination.
* Has a usable pair of spectacle lenses if required for transportation to the site for the initial visit

Exclusion Criteria:

* Is presently participating in any other clinical or research study including eye related clinical or research study.
* Has never worn contact lenses before.
* Has any systemic disease affecting ocular health.
* Has any active ocular pathology or severe insufficiency of lacrimal secretion (moderate to severe dry eyes) that would affect the wearing of contact lenses.
* Is using any systemic or topical medications that will affect a study outcome variable, and/or ocular health.
* Has any known sensitivity to fluorescein dye or products to be used in the study.
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye.
* Has any clinically significant lid or conjunctival abnormalities, active neovascularization or any central corneal scars.
* Is aphakic.
* Has undergone corneal refractive surgery.
* Is pregnant, lactating, or planning a pregnancy at the time of enrollment (by verbal confirmation at the screening visit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-06-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University Eye Center at Ketchum Health, Anaheim, California
  - Clinical Optics Research Lab (CORL) Indiana University School of Optometry, Indiana University, Bloomington, Indiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Lens Then Control Lens: Subjects were randomized to wear the test lens for one week then the control lens for one week.
  Test lens: contact lens
- Control Lens Then Test Lens: Subjects were randomized to wear the control lens for one week then the test lens for one week.
  Control lens: contact lens
Period: First Intervention
Arm/Group | Test Lens Then Control Lens | Control Lens Then Test Lens
Started | 27 | 25
Completed | 27 | 25
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Test Lens Then Control Lens | Control Lens Then Test Lens
Started | 27 | 25
Completed | 27 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Total Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 52
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Lens Centration
Description: Centration: Grade degree of Centration (Optimally Centered, Slightly Decentered (<0.5mm Nasal (N), T (Temporal), S (superior), I (inferior), Extremely Decentered (>0.5mm N T S I)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Test Lens: Subjects were randomized to wear the test lens for one week.
  Test lens: contact lens
- Control Lens: Subjects were randomized to wear the control lens for one week.
  Control lens: contact lens
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 52 | 52
Participants
  Optimal | 17 | 12
  Slightly Decentered | 34 | 39
  Extreme Decentered | 1 | 1

2. Primary Outcome: Number of Participants With Lens Centration
Description: as for outcome 1
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 52 | 52
Participants
  Optimal | 20 | 16
  Slightly Decentered | 31 | 36
  Extreme Decentered | 1 | 0

3. Primary Outcome: Post Blink Movement
Description: Post Blink Movement (Amount of movement to the nearest 0.1mm immediately after the blink)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 52 | 52
millimeters (mm) | 0.25 (0.10) | 0.26 (0.09)

4. Primary Outcome: Post Blink Movement
Description: Post Blink Movement (Amount of movement to the nearest 0.1mm immediately after the blink)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 52 | 52
millimeters (mm) | 0.26 (0.12) | 0.25 (0.12)

5. Primary Outcome: Primary Gaze Lag
Description: Primary Gaze Lag (measured in mm at 0.1mm steps)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 52 | 52
millimeters (mm) | 0.22 (0.12) | 0.25 (0.16)

6. Primary Outcome: Primary Gaze Lag
Description: Primary Gaze Lag (measured in mm at 0.1mm steps)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 52 | 52
millimeters (mm) | 0.23 (0.12) | 0.22 (0.15)

7. Primary Outcome: Up Gaze Lag
Description: Up Gaze Lag (measured in mm at 0.1mm steps)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 52 | 52
millimeters (mm) | 0.28 (0.10) | 0.31 (0.12)

8. Primary Outcome: Up Gaze Lag
Description: Up Gaze Lag (measured in mm at 0.1mm steps)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 52 | 52
millimeters (mm) | 0.28 (0.12) | 0.29 (0.20)

9. Primary Outcome: Push-Up Tightness
Description: Push-Up Tightness (measured in 1% steps where 0% Falls from cornea without lid support, 50% optimum, 100% no movement)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 52 | 52
percentage | 46 (6) | 47 (4)

10. Primary Outcome: Push-Up Tightness
Description: Push-Up Tightness (measured in 1% steps where 0% Falls from cornea without lid support, 50% optimum, 100% no movement)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 52 | 52
percentage | 45 (6) | 48 (9)

11. Primary Outcome: Overall Fit Acceptance
Description: Overall fit acceptance assessed on a scale of 0-4 (0=unacceptable - cant be worn, 1 =Acceptable -Poor/worn under supervision, 2 =Acceptable -Fair, prefer refit, 3 = Acceptable-Good, 4 =Acceptable -Optimum
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 52 | 52
units on a scale | 3.12 (0.39) | 3.08 (0.36)

12. Primary Outcome: Overall Fit Acceptance
Description: as for outcome 11
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 52 | 52
units on a scale | 3.12 (0.41) | 3.13 (0.44)

13. Primary Outcome: Number of Participants With Overall Lens Fit Impression
Description: Overall Lens Fit Impression (2=Reduced movement, unacceptable, 1 = Reduced movement acceptable, 0 - Optimal movement, -1 =Excessive movement acceptable, -2 Excessive movement unacceptable
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 52 | 52
Participants
  Reduced Unacceptable | 0 | 0
  Reduced Acceptable | 7 | 7
  Optimal | 43 | 44
  Excessive Acceptable | 2 | 1
  Excessive Unacceptable | 0 | 0

14. Primary Outcome: Number of Participants With Overall Lens Fit Impression
Description: as for outcome 13
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 52 | 52
Participants
  Reduced Unacceptable | 0 | 1
  Reduced Acceptable | 9 | 9
  Optimal | 41 | 41
  Excessive Acceptable | 2 | 1
  Excessive Unacceptable | 0 | 0

15. Secondary Outcome: Subjective Comfort Rating
Description: Subjective comfort scored 0-10 (0-10 scale, 0=uncomfortable, 10 = comfortable)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 52 | 52
units on a scale | 9.0 (1.2) | 9.4 (0.9)

16. Secondary Outcome: Subjective Comfort Rating
Description: Subjective comfort scored 0-10 (0-10 scale, 0=uncomfortable, 10 = comfortable)
Time Frame: 1-week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 52 | 52
units on a scale | 9.1 (1.1) | 9.1 (1.0)

ADVERSE EVENTS:
Time Frame: From baseline up to 1 week for each intervention, a total of 2 weeks.
Groups:
- Control Lens: Subjects were randomized to wear the test lens for one week.
  Control lens: contact lens
Arm/Group | Test Lens | Control Lens
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT03951610/Prot_SAP_000.pdf